CLINICAL TRIAL: NCT07110909
Title: Does HPV Education Affect Knowledge, Awareness, and Concern?
Brief Title: Impact of HPV Education on Knowledge, Awareness, and Concern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gizem ÇITAK (Other)
Responsible Party: Sponsor-Investigator, Gizem ÇITAK, Assistant Professor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K22.05
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Human Papilloma Virus (HPV)
Keywords: HPV; education; knowledge level; awareness; midwife

STUDY DESIGN:
Intervention Model Description: experimental group: 50; control group: 53
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No HPV Education (No Intervention): Control group without HPV education.
- Experimental (Experimental): Participants received HPV education to increase awareness and prevention of cervical cancer
  Interventions: Other: HPV Education

INTERVENTIONS:
Other: HPV Education — HPV Education
  Arms: Experimental

SUMMARY:
This randomized controlled study is being conducted between January and April 2025 at a Family Health Center in the Black Sea Region with 103 women (intervention group: 50, control group: 53) selected via randomizer.org. Participants complete pre-tests, receive HPV and cervical cancer prevention education, and take post-tests to evaluate the impact of the intervention.

Keywords: HPV, education, knowledge, awareness, midwife.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial aimed at evaluating the impact of educational interventions on HPV awareness, knowledge levels, and concerns among women. The research is being carried out at a Family Health Center in the Black Sea Region between January and April 2025. A total of 103 women have been selected through randomizer.org and assigned to either the intervention group (n=50) or control group (n=53).

Participants are initially assessed using a Personal Information Form, the HPV Knowledge Scale, and the HPV Awareness and Concern Scale. The intervention group receives structured education on HPV and cervical cancer prevention delivered by midwives and healthcare professionals. Post-tests are planned to assess potential changes in the measured variables. The study emphasizes the importance of healthcare-based education in improving public awareness and preventive health behaviors.

Keywords: HPV, education, knowledge, awareness, prevention, midwife, cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman aged 18-49
* Not having received any previous education about HPV
* Volunteering to participate in the study and providing written consent

Exclusion Criteria:

* Having been diagnosed with HPV or being in treatment
* Having previously received information or counselling about HPV
* Refusing or withdrawing from the education and data collection process

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 103 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
HPV Knowledge Increase | 1 week
  The increase in women's knowledge about HPV is measured using an HPV knowledge questionnaire. The questionnaire is scored from 0 to 20 points, with higher scores indicating greater knowledge.

SECONDARY OUTCOMES:
Increasing HPV awareness among women | 1 week
  HPV awareness among women is measured using the HPV Awareness Questionnaire, scored from 0 to 10. Higher scores indicate higher awareness of HPV.

CONTACTS AND LOCATIONS:
Overall Officials: GİZEM ÇITAK, Asist. Prof, Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Tokat Gaziosmanpaşa University Rectorate General Secretariat Taşlıçiftlik Campus, 60250 Tokat/Central, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared because the data include sensitive health information and participants did not consent to data sharing.